CLINICAL TRIAL: NCT05310110
Title: The Impact of Using Muscle Relaxants and Laryngeal Local Anesthetics for Laryngeal Mask Airway (LMA) Insertion on Hemodynamics and Induction Anesthetics Dosage in Elderly
Brief Title: Muscle Relaxants and Laryngeal Local Anesthetics for Laryngeal Mask Airway Insertion Decreasing Propofol in Elderly
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Ting, Hung, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 202200004A3
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia, General
Keywords: Muscle relaxants; Laryngeal local anesthetics; Laryngeal mask airway, Laryngeal Masks, LMA; Propofol; Elderly, Aged
MeSH Terms: conditions — Muscle Hypotonia | interventions — cisatracurium; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10% lidocaine spray and cisatracurium group (Experimental): The subjects received laryngeal local anesthetics (10% lidocaine spray), intravenous cisatracurium 0.12 mg/kg, and propofol before laryngeal mask airway placement. The predetermined dosage of propofol for the first subject is 1 mg/kg.
  Interventions: Drug: 10% lidocaine spray; Drug: Cisatracurium; Drug: Propofol
- 10% lidocaine spray and placebo of cisatracurium group (Experimental): The subjects received laryngeal local anesthetics (10% lidocaine spray), intravenous normal saline as a substitute for cisatracurium, and propofol before laryngeal mask airway placement. The predetermined dosage of propofol for the first subject is 1.25 mg/kg.
  Interventions: Drug: 10% lidocaine spray; Drug: Placebo of cisatracurium; Drug: Propofol
- Placebo of lidocaine spray and cisatracurium group (Experimental): The subjects received normal saline spray as a substitute for laryngeal local anesthetics (10% lidocaine spray), intravenous cisatracurium 0.12 mg/kg, and propofol before laryngeal mask airway placement. The predetermined dosage of propofol for the first subject is 1 mg/kg.
  Interventions: Drug: Placebo of lidocaine spray; Drug: Cisatracurium; Drug: Propofol
- Placebo group (Placebo Comparator): The subjects received normal saline spray as a substitute for laryngeal local anesthetics (10% lidocaine spray), intravenous normal saline as a substitute for cisatracurium, and propofol before laryngeal mask airway placement. The predetermined dosage of propofol for the first subject is 2 mg/kg.
  Interventions: Drug: Placebo of lidocaine spray; Drug: Placebo of cisatracurium; Drug: Propofol

INTERVENTIONS:
Drug: 10% lidocaine spray — 10% lidocaine spray 3 puff for the throat before induction
  Arms: 10% lidocaine spray and cisatracurium group; 10% lidocaine spray and placebo of cisatracurium group
Drug: Placebo of lidocaine spray — Normal saline spray 3 puff for the throat before induction
  Arms: Placebo group; Placebo of lidocaine spray and cisatracurium group
Drug: Cisatracurium — Intravenous cisatracurium 0.12 mg/kg during induction
  Arms: 10% lidocaine spray and cisatracurium group; Placebo of lidocaine spray and cisatracurium group
Drug: Placebo of cisatracurium — Intravenous normal saline during induction
  Arms: 10% lidocaine spray and placebo of cisatracurium group; Placebo group
Drug: Propofol — The dosage of intravenous propofol for the first subjects was predetermined for each arm, and the dosage for the subsequent subjects would be determined according to the response of the previous subjects using the Dixon's up-and-down method with a step size of 0.25 mg/kg. If the subjects had no movement and stable hemodynamic status during and after the laryngeal mask airway (LMA) placement, the predetermined dosage of propofol for the subsequent subject would be decreased by 0.25 mg/kg. On the other hand, if the subjects had obvious movement, failure to LMA placement, and significant hemodynamic changes, the predetermined dosage of propofol for the subsequent subject would be increased by 0.25 mg/kg.

SUMMARY:
Laryngeal mask airway (LMA) is currently the most widely used supraglottic airway device with advantages of simple and fast placement, reduced anesthesia drug use, more stable hemodynamics, and less throat discomfort after anesthesia compared to endotracheal intubation. Some studies claimed the use of muscle relaxants or local anesthetics (sprays or lubricants containing local anesthetics) for the throat before LMA placement can reduce the dosage of induction agents and postoperative throat complications.

In modern society, more and more elderly people undergo elective surgery with the need of general anesthesia. However, they are the more vulnerable population with tendency of greater hemodynamic changes with more induction agent usage. Propofol is one of the most used induction agents which may lead to a drop in blood pressure. The objective of this study is to observe whether the dose of propofol and the changes in hemodynamics can be reduced by using muscle relaxants or laryngeal local anesthetics in elderly who receiving general anesthesia with LMA insertion.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Age: over 65 years
* Elective orthopedic surgery undergo general anesthesia in supine position

Exclusion Criteria:

* Anticipated difficult airway (Mallampati score 3-4), limited mouth opening, intra-oral and pharyngeal pathology
* Risk of pulmonary aspiration of gastric contents (full stomach)
* Obesity (Body mass index > 35)
* Significant lung abnormalities (low lung compliance, high airway resistance, impaired oxygenation)
* Loosening teeth
* Allergic to Cisatracurium or Lidocaine
* Failure in successful LMA insertion after second attempts

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Propofol requirement | one minute after propofol infusion
  The minimal propofol requirement dose was defined as the median effective dose (ED50) of movement or increased mean arterial pressure (MAP) to no movement or stable MAP. The ED50 is the average of the crossover midpoints found during conducting the Dixon's up-and-down method.

SECONDARY OUTCOMES:
Non-invasive blood pressure (NIBP) | 0 minute, 1 minute, 2 minute, 3 minute, 4 minute, 5 minute, 10 minute after LMA placement
  Using the non-invasive blood pressure machine to collect the systolic blood pressure, diastolic blood pressure, and mean arterial pressure
Heart rate (HR) | 0 minute, 1 minute, 2 minute, 3 minute, 4 minute, 5 minute, 10 minute after LMA placement
  Using the electrocardiogram monitor to collect the real-time heart rate
Oxygen saturation (SpO2) | 0 minute, 1 minute, 2 minute, 3 minute, 4 minute, 5 minute, 10 minute after LMA placement
  Using the pulse oximeter to collect the real-time oxygen saturation
Peak pressure (P peak) of the airway | 0 minute after LMA placement
  One of the monitoring parameter demonstrated on the mechanical ventilator
Mean pressure (P mean) of the airway | 0 minute after LMA placement
  One of the monitoring parameter demonstrated on the mechanical ventilator
Ease of jaw opening | Procedure (At the same time of LMA placement)
  A factor for evaluating the condition of LMA insertion
Ease of LMA insertion | Procedure (At the same time of LMA placement)
  A factor for evaluating the condition of LMA insertion
Coughing or gagging | Within 1 minute after LMA placement
  Symptoms which suggest non-optimal condition of LMA insertion
Hiccups | Within 1 minute after LMA placement
  Symptoms which suggest non-optimal condition of LMA insertion
Head or body movement | Within 1 minute after LMA placement
  Symptoms which suggest non-optimal condition of LMA insertion
Laryngospasm | Within 1 minute after LMA placement
  Laryngospasm is defined as airway obstruction with assumption that LMA is correctly placed, which is also a factor for evaluating the condition of LMA insertion
Attempts for LMA insertion | Procedure (At the same time of LMA placement)
  The number of attempts for LMA insertion
Complications | One hour after LMA removal
  Including sore throat, dysphagia, dysphonia

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yung-Tai, MD, Study Chair — Department of Anesthesiology, Chang Gung Memorial Hospital, Linkou Medical Center; Hung Yu-Ting, MD, Principal Investigator — Department of Anesthesiology, Chang Gung Memorial Hospital, Linkou Medical Center
Locations (1):
- Linkup Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No